CLINICAL TRIAL: NCT05298904
Title: Pro-active Genetic Testing in Kidney Transplant Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Girish K. Mour, Principal Investigator, Mayo Clinic
Other Study IDs: 21-009697; NCI-2022-02382 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2022-03-11; First posted 2022-03-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked to provide a blood sample. Participants may be asked to provide an additional research blood sample for biobanking purposes, up to 40mL of blood per subject .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney Transplants: Kidney transplant patients who are within one-year post transplant.
  Interventions: Diagnostic Test: Genetic Health Screen Panel

INTERVENTIONS:
Diagnostic Test: Genetic Health Screen Panel — This panel covers cardiomyopathy genes, and cancer genes. The results of this panel are reported as Positive (pathogenic or likely pathogenic mutation identified in one or more genes) or Negative (no pathogenic/likely pathogenic mutations identified).

SUMMARY:
The purpose of this study is to determine the prevalence of genetic mutations that increase the risk of cancer and other medically actionable diseases in kidney transplant patients and to assess the impact of genetic testing on subsequent surveillance for cancer.

ELIGIBILITY:
Inclusion Criteria:

- Post transplant Kidney and Kidney Pancreas recipients.

Exclusion Criteria:

* Simultaneous Liver Kidney Transplant.
* Simultaneous Heart Kidney Transplant.
* Non renal transplant history.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified internally to Mayo Clinic Arizona via the kidney transplant program within one-year post transplant.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2037-03-01 (Estimated); Study Completion 2038-03-01 (Estimated)

PRIMARY OUTCOMES:
Genetic mutations of cancer | 1 year
  Number of subjects to have genetic mutations of cancer in kidney transplant patients receiving care at Mayo Clinic Arizona

SECONDARY OUTCOMES:
The impact of genetic testing | 1 year
  Current guidelines for cancer screening have limitations, as its mostly age based. Immunosuppression can lead to a increased risk of cancer in the kidney transplant population.
  By utilizing a multi gene panel we'll look for the number subjects with positive findings and see how recommendations of care change vs standard of care as recommended by the National Comprehensive Cancer Network (NCCN). Genetic testing and family history may change the practice regarding cancer screening in subjects undergoing kidney transplant evaluation.
Develop a Biorepository | 1 year
  Create a biorepository based on whole exome sequencing and clinical data for future analysis

OTHER OUTCOMES:
Genetic mutations of cardiomyopathy | 1 year
  Prevalence of genetic mutations for cardiomyopathies in kidney transplant recipients

CONTACTS AND LOCATIONS:
Overall Officials: Girish Mour, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials